CLINICAL TRIAL: NCT03405155
Title: Phase II Study of Adjuvant Nivolumab in Patients With Resected Stage IIB/IIC Melanoma
Brief Title: Nivolumab in Treating Patients With Stage IIB-IIC Melanoma That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.641; JT 11821 (Other: JeffTrial Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over at least 30 minutes on day 1. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; NIVO; Opdivo; ONO-4538

SUMMARY:
This phase II trial studies how well nivolumab works in treating patients with stage IIB-IIC melanoma that can be removed by surgery. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy nivolumab administered in the adjuvant setting in patients with resected stage IIB or stage IIC cutaneous melanoma.

SECONDARY OBJECTIVES:

I. To evaluate and estimate the median duration of overall survival (OS) in stage IIB-IIC melanoma patients.

II. To evaluate and estimate the median duration of distant metastases-free survival (DMFS) in stage IIB-IIC melanoma patients.

III. To assess safety and toxicity using Common Terminology Criteria for Adverse Events (CTCAE) version (V)5.

IV. To assess quality of life using the Functional Assessment of Cancer Therapy-Melanoma (FACT-M) quality of life instrument.

TERTIARY OBJECTIVES:

I. To assess and compare clinical, histological, immunological and molecular panels as prognostic and predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completely resected (as per standard of care) melanoma of cutaneous origin in order to be eligible for this study; patients must be classified as stage IIB or IIC cutaneous melanoma using the American Joint Committee on Cancer eighth edition; patients with melanoma of mucosal or other non-cutaneous origin are not eligible; patients with melanoma of ocular origin are not eligible
* Patients must have a negative sentinel lymph node biopsy or undergo a failed attempt at sentinel lymph node biopsy including lymphoscintography which fails to show a sentinel lymph node from the melanoma primary site
* Patients must have systemic cross-sectional imaging (positron emission tomography [PET]/computed tomography [CT] or CT of chest, abdomen, and pelvis) which shows no evidence of metastatic disease
* Patient must be able to comprehend and sign a written informed consent and be willing to comply with all study procedures
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1,500 microliter (mcL)
* Platelets >= 100,000/mcL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) (except Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) and alkaline phosphatase =< 2 x institutional upper limit of normal (IULN)
* Serum creatinine =< 1.5xULN OR measured or calculated creatinine clearance >= 60 mL/min
* Patients known to be human immunodeficiency virus (HIV) positive are eligible if they meet the following criteria within 30 days prior to registration: stable and adequate CD4 counts (>= 350 mm^3), and serum HIV viral load of < 25,000 IU/ml; patients may be on or off anti-viral therapy so long as they meet the CD4 count criteria
* Women of childbearing potential must have a negative urine or serum pregnancy test within 28 days prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method for the course of the study through 120 days after the last dose of study medication; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures; patients must not be pregnant or nursing
* Therapy must be initiated within 120 days of surgical resection of the sentinel lymph nodes and within 6 months of initial diagnosis.
* Patients must be willing to have archived tumor specimens utilized for correlative studies if available
* Patients must not have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection prior to registration

Exclusion Criteria:

* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, lobular carcinoma of the breast in situ, atypical melanocytic hyperplasia or melanoma in situ, adequately treated stage I or II cancer (including multiple primary melanomas) from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Current immunosuppressive therapy including > 10 mg/day of prednisone within 14 days of enrollment is not permitted; inhaled or topical steroids, and adrenal replacement steroid doses =< 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients must not have a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients must not have received live vaccines within 42 days prior to registration; examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine; seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Patients must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the trial results, interfere with the patient's participation for the full duration of the trial, or indicate that participation in the trial is not in the patient's best interests, in the opinion of the treating investigator
* Patients must not be pregnant or lactating
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) is not permitted
* Treatment with any investigational agent within 14 days of first administration of study treatment is not permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival | Up to 24 months
  Will be estimated by the Kaplan-Meier method. The corresponding median survival times (with 90% confidence limits) will be determined, as will the cumulative percentage of patients remaining progression-free / alive at selected time points after initial treatment (e.g., 6, 12, and 18 months).

SECONDARY OUTCOMES:
Median duration of overall survival | Up to 24 months
  Will be estimated by the Kaplan-Meier method. The corresponding median survival times (with 90% confidence limits) will be determined, as will the cumulative percentage of patients remaining progression-free/alive at selected time points after initial treatment (e.g., 6, 12, and 18 months).
Median duration of distant metastases-free survival | Up to 24 months
  Will be estimated by the Kaplan-Meier method. The corresponding median survival times (with 90% confidence limits) will be determined, as will the cumulative percentage of patients remaining progression-free/alive at selected time points after initial treatment (e.g., 6, 12, and 18 months).
Number of Adverse Events | Up to 24 months
  Will be assessed by Common Terminology Criteria for Adverse Events version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Takami Sato, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (4):
- United States (4):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Columbia University, New York, New York
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/